CLINICAL TRIAL: NCT02550132
Title: Neuromechanical Response to Spinal Manipulation Therapy: Effects of a Constant Rate of Force Application
Brief Title: The Role of the Rate of Force Application in Responses to Spinal Manipulation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Fondation Chiropratique du Québec (Other)
Responsible Party: Principal Investigator, Martin Descarreaux, Dr Martin Descarreaux DC, PhD, Université du Québec à Trois-Rivières
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UQTR-2013-SMTrate
Record Dates: First submitted 2015-09-08; First posted 2015-09-15 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Spinal Manipulation
Keywords: electromyography; biomechanical phenomena; dose-response relationship; musculoskeletal manipulations; spinal manipulation
MeSH Terms: interventions — Manipulation, Spinal; Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants (Experimental): All volunteers will participate in an experimental session. Participants will be delivered four different spinal manipulations (SMT) at T7 with a rate of force application of about 2200 Newtons/seconds and a preload force of 25 Newtons (N). SMTs will differed in their time to peak force (ms) and peak force (N), respectively fixed as follow for each applied SMT: (1)57 ms / 150 N, (2)80 ms / 200 N, (3)102 ms / 250 N and (4)125 ms / 300 N.
  Interventions: Procedure: Spinal manipulation; Device: Apparatus used to deliver spinal manipulations

INTERVENTIONS:
Procedure: Spinal manipulation — Participants will lie down during the 45-minute experimental session. Vertebral displacements (cm) and muscle response amplitude (RMS value) will be recorded through kinematic markers (on T6, T7 and T8 spinous processes) and surface electromyography electrodes (on the left and right erector spinae at T6 and T8 vertebra level). Each SMT (4 per participant) will be delivered at T7 transverse processes by an apparatus. Responses during the thrust phase (duration equal to twice the time to peak force) and after the thrust (1,5s duration) will be compared between SMTs.
  Other Names: Manual therapy
Device: Apparatus used to deliver spinal manipulations — An apparatus using a servo-controlled linear actuator motor (Linear Motor Series P01-48x360, LinMot Inc., Switzerland) will be used to deliver spinal manipulations.

SUMMARY:
The objective of the present study is to determine if spinal manipulations with a constant rate of force application but with different peak force and time to peak force lead to similar responses in healthy adults.

DETAILED DESCRIPTION:
Although there are indirect evidences that the rate of force application modulates neuromuscular responses to spinal manipulation therapy (SMT) through peak force or thrust duration modulations, such an assumption remains to be confirmed. Therefore, the objective of the present study was to determine if different SMT force-time profiles where a constant rate of force application would be maintained (through the modulation of the peak force and the time to peak force) lead to similar neuromechanical responses. Based on the available data relative to the effect of SMT biomechanical parameters modulation, it was hypothesized that neuromuscular responses would be similar across SMT force-time profiles, while vertebral displacements would increase as SMT peak force increases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult

Exclusion Criteria:

* Thoracic or lumbar pain
* History of back trauma or surgery
* Severe osteoarthritis
* Inflammatory arthritis
* Vascular conditions
* Contraindication to the use of SMT

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Descarreaux, DC, PhD, Principal Investigator — Université du Québec à Trois-Rivières

REFERENCES:
- [Derived] Nougarou F, Page I, Loranger M, Dugas C, Descarreaux M. Neuromechanical response to spinal manipulation therapy: effects of a constant rate of force application. BMC Complement Altern Med. 2016 Jun 2;16:161. doi: 10.1186/s12906-016-1153-6. PMID 27249939

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.76 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Region of Enrollment [Number; unit: participants]
  Canada | 25

OUTCOME MEASURES:

1. Primary Outcome: Left T6 Normalized Root Mean Square (RMS) Value
Description: Normalized amplitude (RMS) of surface electromyography response. The normalisation was achieved by dividing the obtained RMS by the RMS value before thrust application.
Time Frame: During the 150N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 3.72 (0.68)

2. Primary Outcome: Left T8 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 150N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 2.83 (0.30)

3. Primary Outcome: Right T6 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 150N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 3.03 (0.35)

4. Primary Outcome: Right T8 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 150N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 3.51 (0.84)

5. Primary Outcome: Left T6 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 200N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 4.75 (0.76)

6. Primary Outcome: Left T8 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 200N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 4.12 (0.50)

7. Primary Outcome: Right T6 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 200N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 3.13 (0.33)

8. Primary Outcome: Right T8 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 200N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 3.46 (0.41)

9. Primary Outcome: Left T6 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 250N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 4.92 (0.91)

10. Primary Outcome: Left T8 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 250N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 4.03 (0.52)

11. Primary Outcome: Right T6 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 250N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 3.40 (0.40)

12. Primary Outcome: Right T8 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 250N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 3.57 (0.55)

13. Primary Outcome: Left T6 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 300N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 4.17 (0.53)

14. Primary Outcome: Left T8 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 300N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 4.80 (0.88)

15. Primary Outcome: Right T6 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 300N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 3.87 (0.64)

16. Primary Outcome: Right T8 Normalized Root Mean Square (RMS) Value
Description: as for outcome 1
Time Frame: During the 300N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Participants
Number analyzed (Participants) | 25
ratio | 3.79 (0.49)

17. Primary Outcome: Vertebral Displacement of the Sixth Thoracic Vertebra
Description: Absolute posterior to anterior vertebral displacement during the spinal manipulation in centimeter
Time Frame: During the 150N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: cm
Arm/Group | Participants
Number analyzed (Participants) | 25
cm | 0.81 (0.04)

18. Primary Outcome: Vertebral Displacement of the Seventh Thoracic Vertebra
Description: Absolute posterior to anterior vertebral displacement during the spinal manipulation in centimeter
Time Frame: During the 150N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: cm
Arm/Group | Participants
Number analyzed (Participants) | 25
cm | 1.01 (0.03)

19. Primary Outcome: Vertebral Displacement of the Eighth Thoracic Vertebra
Description: Absolute posterior to anterior vertebral displacement during the spinal manipulation in centimeter
Time Frame: During the 150N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: cm
Arm/Group | Participants
Number analyzed (Participants) | 25
cm | 0.76 (0.04)

20. Primary Outcome: Vertebral Displacement of the Sixth Thoracic Vertebra
Description: Absolute posterior to anterior vertebral displacement during the spinal manipulation in centimeter
Time Frame: During the 200N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: cm
Arm/Group | Participants
Number analyzed (Participants) | 25
cm | 1.18 (0.07)

21. Primary Outcome: Vertebral Displacement of the Seventh Thoracic Vertebra
Description: Absolute posterior to anterior vertebral displacement during the spinal manipulation in centimeter
Time Frame: During the 200N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: cm
Arm/Group | Participants
Number analyzed (Participants) | 25
cm | 1.32 (0.06)

22. Primary Outcome: Vertebral Displacement of the Eighth Thoracic Vertebra
Description: Absolute posterior to anterior vertebral displacement during the spinal manipulation in centimeter
Time Frame: During the 200N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: cm
Arm/Group | Participants
Number analyzed (Participants) | 25
cm | 1.10 (0.05)

23. Primary Outcome: Vertebral Displacement of the Sixth Thoracic Vertebra
Description: Absolute posterior to anterior vertebral displacement during the spinal manipulation in centimeter
Time Frame: During the 250N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: cm
Arm/Group | Participants
Number analyzed (Participants) | 25
cm | 1.48 (0.06)

24. Primary Outcome: Vertebral Displacement of the Seventh Thoracic Vertebra
Description: Absolute posterior to anterior vertebral displacement during the spinal manipulation in centimeter
Time Frame: During the 250N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: cm
Arm/Group | Participants
Number analyzed (Participants) | 25
cm | 1.69 (0.05)

25. Primary Outcome: Vertebral Displacement of the Eighth Thoracic Vertebra
Description: Absolute posterior to anterior vertebral displacement during the spinal manipulation in centimeter
Time Frame: During the 250N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: cm
Arm/Group | Participants
Number analyzed (Participants) | 25
cm | 1.40 (0.05)

26. Primary Outcome: Vertebral Displacement of the Sixth Thoracic Vertebra
Description: Absolute posterior to anterior vertebral displacement during the spinal manipulation in centimeter
Time Frame: During the 300N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: cm
Arm/Group | Participants
Number analyzed (Participants) | 25
cm | 1.74 (0.09)

27. Primary Outcome: Vertebral Displacement of the Seventh Thoracic Vertebra
Description: Absolute posterior to anterior vertebral displacement during the spinal manipulation in centimeter
Time Frame: During the 300N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: cm
Arm/Group | Participants
Number analyzed (Participants) | 25
cm | 1.40 (0.08)

28. Primary Outcome: Vertebral Displacement of the Eighth Thoracic Vertebra
Description: Absolute posterior to anterior vertebral displacement during the spinal manipulation in centimeter
Time Frame: During the 300N spinal manipulation procedure, assessed up to 2 seconds following thrust onset
Measure: Mean (Standard Error); unit: cm
Arm/Group | Participants
Number analyzed (Participants) | 25
cm | 1.70 (0.07)

ADVERSE EVENTS:
Time Frame: Adverse event were collected during the 45 min experimental session
Description: Participants were invited to express their pain or discomfort during the experimental session.
Arm/Group | Participants
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No